CLINICAL TRIAL: NCT04273776
Title: A Comparison of the Physiological and Behavioral Effects of Suvorexant and Zolpidem in Healthy Volunteers: A Randomized, Double-blind, Placebo Controlled Study
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Walter Reed Army Institute of Research (WRAIR) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Other
Other Study IDs: WRAIR #2492
Record Dates: First submitted 2020-02-14; First posted 2020-02-18 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Performance Enhancing Product Use
MeSH Terms: interventions — suvorexant; Zolpidem

STUDY DESIGN:
Intervention Model Description: Randomization will occur at the level of the study session such that all volunteers participating in the same session will be "blocked" together (i.e., assigned the same condition).
Who Masked: Participant, Investigator
Masking Description: Study sessions will be randomized prior to the study (e.g. Session 1 = placebo, Session 2 = zolpidem, etc.) and volunteers will be assigned a session (treatment group) when they are scheduled for their enrollment visit (Day 1). The randomization schedule will be generated using a random number generator by a person who is not involved in data collection prior to commencement of the study, with the following qualification (hence "pseudo-random"): that all volunteers participating in the same session be randomized or "blocked" together (i.e., assigned the same condition). This will help ensure double-blinding since it may be obvious to volunteers and staff within the same session if some volunteers receive placebo whereas others receive active drug. To help maintain confidentiality, each participant will also be given a unique numerical identifier (e.g., 01-120).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Suvorexant Arm (Active Comparator): 10 mg of Suvorexant
  Interventions: Drug: Suvorexant 10 mg; Drug: Placebos
- Zolpidem Arm (Active Comparator): 5 mg of Zolpidem
  Interventions: Drug: Zolpidem; Drug: Placebos
- Placebo (Placebo Comparator): 10mg of Avicel
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Suvorexant 10 mg — 10 mg of suvorexant
  Arms: Suvorexant Arm
Drug: Zolpidem — 5 mg of zolpidem
  Arms: Zolpidem Arm
Drug: Placebos — Avicel

SUMMARY:
The primary objective of this study is to evaluate two pharmacotherapeutic approaches to sleep induction, both of which have been shown to be effective hypnotics, but may have unique side effect profiles. These profiles may have markedly different impacts on performance in a military setting. In this randomized, double-blind, placebo controlled study, the side effects of these drugs will be compared - suvorexant, a dual orexin receptor antagonist and zolpidem, a non-benzodiazepine gamma-aminobutyric acid (GABA) A agonist - in healthy controls comparable in age and gender to the target military population.

ELIGIBILITY:
Inclusion Criteria

Healthy males and non-pregnant, non-lactating female volunteers must be between the ages of 18 and 39

* learned English as a first language (inclusive)*.
* To be included in the study, volunteers will have to pass a "Volunteer Comprehension Assessment" with a score of 80% or greater. A maximum of two attempts is permitted. See section 5.7 for details.
* Females of child-bearing potential must be on some form of birth control, if sexually active (e.g., oral contraceptive, condom, intrauterine device, etc.)

  * Volunteers must have learned English as their first language. This is because there are cognitive tests administered during the study that require a mastery of the English language.

Exclusion Criteria

* Self-reported habitual nightly sleep amounts outside the target range of approximately 6-9 hours (i.e., less than 6 hours per night or more than 9 hours per night, on average) (Post-consent Checklist).
* Any use of prescription or over-the-counter sleep aids during the 3-month period prior to screening determined by the examining study medical investigator to be indicative of a potential sleep disorder (e.g., use of a sleep aid for several nights following travel across multiple time zones would not necessarily constitute evidence of a sleep disorder).
* Self-reported nighttime lights-out times earlier than 2000 or later than 0100 during weeknights (Sunday through Thursday) (Post-consent Checklist)
* Self-reported morning wake-up times earlier than 0500 or later than 0900 during weekdays (Monday through Friday) (Post-consent Checklist)
* Self-reported habitual napping (> 3 times a week) in conjunction with normal sleep habits (Post-consent Checklist).
* Self-reported symptoms suggestive of a sleep disorder (including but not limited to insomnia, narcolepsy, sleep disordered breathing/sleep apnea, idiopathic hypersomnia, restless leg syndrome, parasomnias, REM behavior disorder, etc.) (Post-Consent Checklist, Medical History/Exam form; Berlin Questionnaire); history of a sleep disorder (Medical History and Examination) or evidence of such from a prior polysomnographic assessment.
* Objective evidence of narcolepsy + cataplexy using the Ullanlinna Narcolepsy Scale
* Objective evidence of insomnia using the Insomnia Severity Index.
* STATE TRAIT ANXIETY INVENTORY - TRAIT (STAI-T) - Scores above 40.
* MORNING-EVENINGNESS QUESTIONNAIRE -Scores lower than 31 or greater than 69.
* Self-reported caffeine use in excess of 400 mg (e.g., approximately 8 caffeinated sodas or approximately 20 ounces of brewed coffee) per day on average (Post-consent Checklist)
* History of neurologic disorder (including but not limited to epilepsy or another seizure disorder, amnesia, hydrocephalus, Parkinson's disease, MS) (Medical History and Examination form). An infrequent or resolved single neurological event (e.g., childhood seizure, rare sporadic migraine headaches, resolved meningeal infection with no sequelae) may be deemed non-exclusionary at the discretion of the examining study medical investigator.
* Score of 14 or above on the Beck Depression Inventory (BDI form)
* History of cardiovascular disease (including but not limited to arrhythmias, valvular heart disease, congestive heart failure, history of myocardial infarction) (Medical History/Exam form)
* Underlying acute or chronic pulmonary disease requiring daily inhaler use (Medical History /Exam form)
* Kidney disease or significant kidney abnormalities (Medical History/Exam form, laboratory results) as determined by examining study medical investigator.
* Liver disease or significant liver abnormalities (Medical History/Exam form, laboratory results) as determined by examining study medical investigator.
* Self-reported history of psychiatric disorder requiring hospitalization or psychiatric medication for more than 6 months (Medical History/Exam form)
* Self-reported or suspected use of products or drugs that cannot be safely discontinued during in-laboratory phases, to be determined on a case-by-case basis by the examining study medical investigator (Medical History/Exam form).
* Self-reported or suspected heavy alcohol use (minimum limit to define heavy alcohol use is 14 drinks per week or as determined by the examining study medical investigator).
* Self-reported or suspected regular nicotine use (or addiction) (defined as more than 1 cigarette or equivalent per week) within the last 1 year.
* Self-reported or suspected current use of other illicit drugs (including but not limited to benzodiazepines, amphetamines, cocaine, marijuana) (Medical History/Exam form)

Positive urine pregnancy result

* Positive salivary alcohol screening result
* Self-reported or suspected current breast-feeding or collecting breast-milk (Medical History/Exam form)
* Resting blood pressure above 140/90 or resting pulse > 110 beats per minute (Medical History/Exam form) Note that if a repeat measurement is within range, volunteer will not be excluded.
* BMI ≥ 30 (Obese Class I or greater) (Medical History/Exam form)
* Clinically significant values (as determined by the reviewing study medical investigator and the table below) for any hematology or chemistry parameter included in the screening bloodwork.
* Positive urine nicotine/cotinine result during screening visit (NicCheckTM I test strip results)
* Positive urine drug screen result
* Inability to read and sign consent
* Failure to obtain required approved official leave to participate
* Presence of features that may increase risk and/or discomfort during the cold pressor task. These include: past cramp attacks or blackouts, chilblains, open skin wounds, fracture of the hands, and skin and peripheral vascular diseases (to include but not limited to Raynaud's disease.
* As prisoners will not be recruited and are not eligible for participation in this study, any participant that becomes incarcerated during Phase 1 will result in termination from the study.

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2019-12-01 (Actual); Primary Completion 2024-11-21 (Actual); Study Completion 2025-12-12 (Estimated)

PRIMARY OUTCOMES:
consolidation of episodic memory | 5 days
  presentation of word lists
psychomotor vigilance test | 4 days
  measures reaction time

CONTACTS AND LOCATIONS:
Locations (1):
- Walter Reed Army Institute of Research, Silver Spring, Maryland, United States

IPD SHARING:
Plan to Share IPD: No